CLINICAL TRIAL: NCT04927715
Title: FDNC5 Genetic Polymorphism in Patients With Peripartum Cardiomyopathy
Brief Title: Irisin Expression and Gene Polymorphism With Peripartum Cardiomyopathy.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ahmed Altaher, clinical professor, Sohag University
Other Study IDs: Soh-Med-21-02-26
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Peripartum Cardiomyopathy
Keywords: Peripartum Cardiomyopathy, Irisin
MeSH Terms: conditions — Peripartum Cardiomyopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diseased: Females with peripartum cardiomyopathy
- Control: Healthy females

SUMMARY:
this is an observertional study aimed at Study the association between the level of irisin expression and (Fibronectin Type III Domain Containing 5 (FDNC5) gene polymorphism in female patients with peripartum cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* This study will include females aged between 18 and 45 years old who have been diagnosed and treated clinically for peripartum cardiomyopathy

Exclusion Criteria:

* Age less than 18 or more than 45 year old
* females with dilated cardiomyopathy due to other etiology or outside the time frame of occurrence of peripartum cardiomyopathy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — the studied disease peripartum cardiomyopathy is female specific
Study Population: females who have been diagnosed and treated clinically for peripartum cardiomyopathy in our center in sohag university hospital
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Irisin level | 4 months
  detect the serum level of irisin hormone by ELIZA in nanogram/decilitre(ng/dl)
FNDC5 Genotyping | 4 months
  whether homogenetic or heterogenetic

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag uniersity hosoital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided